CLINICAL TRIAL: NCT02148315
Title: School Gardens and Physical Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: RWFJ 69550
Record Dates: First submitted 2014-05-23; First posted 2014-05-28 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2014-05

CONDITIONS: Physical Activity
Keywords: physical activity; children; school; garden
MeSH Terms: conditions — Motor Activity | interventions — Gardens

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- garden intervention (Experimental): garden kit and access to garden-based lessons
  Interventions: Behavioral: garden
- no garden (No Intervention): control - receives garden and lessons at end of study

INTERVENTIONS:
Behavioral: garden
  Arms: garden intervention

SUMMARY:
The purpose of this study is to determine whether school gardens affect children's physical activity.

DETAILED DESCRIPTION:
New York State schools were randomly assigned to receive school gardens and associated curriculum or to serve on the wait list control group that received gardens and curriculum at the end of the 2-year study. Baseline data were collected in Fall 2011. Garden interventions began in Spring 2012. Follow-up data were collected at 6, 12, 18 months following baseline data collection.

ELIGIBILITY:
Inclusion Criteria:

* schools had at least 50% of enrolled children qualifying for free + reduced price meals (FRPM)
* schools did not already have a school garden

Exclusion Criteria:

-

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 234 (Actual)
Dates: Start 2011-08; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
change in physical activity | change from baseline to follow-ups at 6, 12, 18 months
  Physical activity was measured using a survey measure, accelerometry, and direct observation.

SECONDARY OUTCOMES:
change in time spent outdoors | baseline to follow-ups at 6, 12, 18 months
  Time spent outdoors was measured by lux using accelerometry

CONTACTS AND LOCATIONS:
Overall Officials: Nancy M Wells, PhD, Principal Investigator — Cornell University
Locations (1):
- Schools in New York State, Ithaca, New York, United States

REFERENCES:
- [Derived] Wells NM, Myers BM, Henderson CR Jr. Study protocol: effects of school gardens on children's physical activity. Arch Public Health. 2014 Dec 8;72(1):43. doi: 10.1186/2049-3258-72-43. eCollection 2014. PMID 25671113
- [Derived] Wells NM, Myers BM, Henderson CR Jr. School gardens and physical activity: a randomized controlled trial of low-income elementary schools. Prev Med. 2014 Dec;69 Suppl 1:S27-33. doi: 10.1016/j.ypmed.2014.10.012. Epub 2014 Oct 16. PMID 25456803
- See also: Active Living Research, Robert Wood Johnson Foundation — http://activelivingresearch.org/